CLINICAL TRIAL: NCT00846534
Title: The Assessment of Oxidative Stress Markers and the Development of Atrial Fibrillation After Cardiac Surgery
Acronym: POAF
Status: Terminated | Type: Observational
Why Stopped: Insufficient patient volume
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Samuel C. Dudley, Professor, University of Illinois at Chicago
Other Study IDs: 2007-0916
Record Dates: First submitted 2009-01-14; First posted 2009-02-18 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Atrial Fibrillation
Keywords: Oxidative stress markers; Cardiac surgery; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Approximately 10- 15 ml of blood will be drawn from subjects. Blood samples will be separated into plasma and serum to measure the oxidative stress markers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post operative atrial fibrillation: To evaluate the ability of oxidative stress markers to predict postoperative atrial fibrillation in subjects undergoing cardiac surgery.

SUMMARY:
The purpose of the investigators study is to investigate the correlation between naturally occurring chemicals, called reactive oxygen species (ROS), in the blood of human patients and the development of an abnormal heart rhythm, known as atrial fibrillation (AF). The development of atrial fibrillation is associated with increased medical problems like stroke. Many factors seem to cause the development of AF, and this rhythm occurs frequently after open heart surgery. When patients develop AF after cardiac surgery they are at increased risk for cognitive changes, infections, the development of kidney failure, and increased length of hospitalization. ROS are chemicals in blood and tissues that tend to cause microscopic blood vessel and heart damage. These chemicals occur naturally as the result of chemical reactions that occur in states of stress and inflammation, like tissue trauma and as the result of smoking. Patients who undergo cardiac surgery may have higher levels of ROS because of their underlying medical conditions. In addition, the organized tissue trauma that occurs in the setting of surgery may serve to increase ROS levels further. In turn, the higher ROS levels may put patients at even higher risk for the development of AF. The investigators believe that increased levels of ROS may help potentiate a patient's development of AF. Accordingly the investigators aim to measure ROS levels before and after surgery to see if there are particular levels that predict the development of this abnormal heart rhythm. By developing a better knowledge of the relationship between ROS and AF, the investigators hope to better understand another possible method of detecting patients who are at the highest risk of developing AF before it occurs after surgery. If these patients are better identified, this may eventually lead to medical treatment to prevent AF; and hopefully this will result in a decrease of the malicious effects that result from developing this abnormal heart rhythm.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is a common occurrence after cardiac surgery. This arrhythmia is reported to occur in up to 40% of patients following coronary bypass graft (CABG) surgery. The incidence of AF is even higher in patients who have undergone both CABG and valvular surgery during the same operation. In cardiac surgery patients, the occurrence of atrial fibrillation post-operatively lengthens hospitalization and adds to postoperative complications like renal dysfunction, infection, and cognitive defects. Postoperative AF is a known major risk factor for the development of stroke after cardiac surgery. Additionally, there is data to suggest that the development of AF after cardiac surgery is related to both reduced survival after CABG, and this dysrhythmia may also serve as an independent predictor of long-term mortality. Many studies have investigated the role of prophylactic pharmacological therapy to prevent post-operative AF after cardiac surgery. Despite this, the complete pathogenesis of AF in the post-cardiac surgery population remains unknown, is likely to be multifactorial, and includes clinical, structural, and biochemical risk factors.

Biochemical risk factors such as inflammation and elevated markers of oxidative stress seem to be related to the development of AF. Also, It has been shown that AF is associated with decreased activity of nitric oxide synthases. Elevated C-reactive protein (CRP), a common marker of inflammation, has been shown to be associated with chronic AF at one year follow up. Additionally, elevated CRP levels drawn just prior to electrical cardioversion have been found to predict the development of recurrent AF after cardioversion. This relationship between this elevated marker of inflammation - CRP - and AF has been found to be independent of clinical risk factors for the development of AF, such as age, diabetes, and left ventricular function. Inflammation is a known source of oxidative stress at the cellular level; and it has been proposed that both inflammation and oxidative stress play a role in electrical remodeling of the atria, which promotes perpetuation of AF. Moreover, it has been proposed that CRP levels may directly reflect the condition of increased oxidative stress.

Oxidative Stress and Arrhythmia:

The association between AF and arrhythmias has been suggested by an array of evidence. Moreover, the pathogenesis likely involves both changes in the atrial architecture, such as dilation and fibrosis, and alterations in the electrophysiological substrate of atrial tissue. Oxidative stress markers are believed to be involved in remodeling of the atrial electrophysiological substrate.

Recently, a correlation between AF and oxidative stress markers has been established. In one study, a correlation between the oxidative stress markers reduced glutathione, cysteine, and derivatives of reduced oxidative metabolites has been found. Although the relationship between AF and oxidative stress remains unclear, it is known from this human population study that oxidative stress markers are elevated in those with persistent AF. This relationship holds true even after controlling for conditions that promote oxidative stress: hypertension, smoking, and congestive heart failure. It has also been shown that atrial tachycardias are associated with increased hydroxyl radicals and peroxynitrite. These species are believed to cause myofibril damage and reduced myofibrillar creatine kinase activity in those with chronic AF. Similarly, superoxide free radicals were shown to be elevated in the porcine heart left atrial appendage when subjected to rapid atrial pacing and AF. Of further interest in this study by Dudley et al., was the role of an NADPH oxidase inhibitor, apocynin, in its ability to reduce superoxide production. This suggests that the NADPH oxidase plays a prominent role in the development of reactive oxidative species. In turn, such reactive oxidative species are thought to be related to inflammation and atrial electrical remodeling.

It is believed that electrical remodeling leads to changes such as shortening of the effective refractory period (ERP), loss of rate adaptation of the refractory period, and prolonged atrial conduction. Rapid atrial conduction likely results in increased calcium (Ca2+) accumulation. This causes decreased inward L-type Ca2+ current (ICa), resulting in a shorter action potential duration (APD). Additional cellular mechanisms may include inactivation of the fast sodium current (INa) at more positive membrane potentials, and increased inward potassium rectifier (IK1) and acetylcholine dependent potassium currents (IKAch). Though these currents logically oppose one another, the net effect is that of increased repolarization heterogenicity and shortened APD. Moreover, experimental models have shown that rapid atrial pacing leads to decreased ERP and reduced of L-type Ca2+ channel and transient outward K+ ion currents. Shortening of the ERP leads to decreased conduction wavelengths, and shortened wavelengths have been proposed to increase the propensity for the development of AF because they reduce the mass of atrial tissue required to sustain reentry circuits.

Given the changes above, it has been postulated that intracellular calcium overload as a result of AF is a trigger for electrical remodeling in AF. Nevertheless, further studies have demonstrated that blockade of L-type calcium channels alone with verapamil in canine hearts is not sufficient to prevent atrial electrical remodeling. Additional triggering mechanisms may include oxidative stress and inflammation. Simvastatin, a drug that has both anti-oxidant and anti-inflammatory properties has been shown to attenuate the development of AF from tachycardia induced atrial remodeling in dogs. More specific evidence of ion channel remodeling from free radicals was proved by Caouette et al. who showed that addition of hydrogen peroxide directly delayed ultra-rapid rectifier potassium currents in the Chinese Hamster Ovary cell line. These changes are mediated by Kv1.5 gene expression, which accounts for voltage-gated potassium repolarization currents that are similarly expressed in human atrial and ventricular myocytes. Further ion channel studies have demonstrated that lipid peroxidation causes Na+ channel dysfunction in cultured atrial myocytes when exposed to the oxidizing agent tert-butyl-hydroperoxide . Additionally, it is believed that reactive oxidative species may promote respiratory chain dysfunction in atrial myocytes by way of mitochondrial DNA damage.

In summary, the relationship between oxidative stress and atrial fibrillation is complex and incompletely understood on the molecular level. Nevertheless, it is clear that this relationship does exist, and therefore serves as a potential focus for medical therapy. In fact, Carnes et al. clearly demonstrated that using ascorbate perioperatively to blunt the effects of oxidative stress results in both decreased peroxynitrite formation and a lower incidence of AF after CABG. Therefore, investigators propose to do more work in this arena to better elucidate the relationship of oxidative stress and AF.

Oxidative Stress Markers in the Research Setting:

Cardiac surgery leads to high oxidative stress and inflammation and is associated with postoperative AF. This is the ideal situation in which to better define oxidative stress markers and their correlation with AF. There are several ways to measure oxidative stress in humans. A minimally invasive method is the measurement of lipid peroxides (derivatives of reactive oxygen metabolites, dROMs) and oxidized and reduced thiol ratios. Glutathione is an important water-phase antioxidant and essential cofactor for antioxidant enzymes. It provides protection endogenous oxygen radicals. Since glutathione can exist in oxidized and reduced forms, it can serve as a buffer for increased oxidative stress. Moreover, the relative amounts of these two forms are a reflection of the oxidative state of humans. This balance can be measured out of blood. Measurement of this ratio has been validated by Neuman et al. and is known to be associated with AF. Additionally, these measurements have been validated in states that are thought to increase oxidative stress, such as diabetes, older age, and cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Sinus rhythm at the time of enrollment as documented by ECG, telemetry, or Holter monitoring
* Scheduled for an open heart surgery
* Able to provide informed consent

Exclusion Criteria:

* Systemic inflammatory diseases (e.g., collagen vascular diseases, infections)
* Malignant neoplasms
* Hyperthyroidism
* Uncontrolled hypertension (blood pressure > 180/100 at rest) on medications
* An illness that might result in death within 1 year
* Implanted devices for designed for active management of atrial arrhythmias by pacing or defibrillation
* Current illicit drug use
* Current ethanol abuse
* Presence of paroxysmal, persistent, or permanent atrial fibrillation at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of this study is all patients who will undergo cardiac surgery. There is no particular age range, but subjects less than 18 years of age will be omitted because of the rarity of AF in this population. The target number of subjects will be 100.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Baseline of oxidative stress markers prior to subjects undergoing cardiac surgery | up to 24 hours pre-op
To evaluate the ability of oxidative stress markers to predict postoperative atrial fibrillation in subjects undergoing cardiac surgery | Day 1 post-op
To evaluate the ability of oxidative stress markers to predict postoperative atrial fibrillation in subjects undergoing cardiac surgery | When develop Atrial Fibrillation or upon discharge from hospital, usually within 1 week post-op

CONTACTS AND LOCATIONS:
Overall Officials: Samuel C Dudley, MD. PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois